CLINICAL TRIAL: NCT06489405
Title: The Effect of Hortıcultural Practices on Internet Addiction, Social Skills and Stress Levels in Children
Brief Title: Horticultural Practices for Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sultan Ayaz Alkaya, Prof. Dr., Faculty of nursing, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-705930
Record Dates: First submitted 2024-06-26; First posted 2024-07-05 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Internet Addiction Level; Perceived Stres Level; Social Skill Level
Keywords: horticultural practices; internet addiction; perceived stres; social skill
MeSH Terms: conditions — Internet Addiction Disorder; Social Skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Horticultural practices (Experimental): Horticultural practices, consisting of 6 sessions with a one-week interval,was applied face to face to this intervention group. Each session lasted approximately 60 minutes.
  Interventions: Other: Horticultural practices
- Control (No Intervention): No intervention has been made.

INTERVENTIONS:
Other: Horticultural practices — The first week of the program was 'Getting to know horticultural practices', the second week was 'Painting pots', the third week was 'Planting vegetable seedlings', the fourth week was 'Preparing compost', the fifth week was 'Making pressed flowers' and the sixth week was 'Harvesting vegetables'.
  Arms: Horticultural practices

SUMMARY:
The study was conducted with a parallel group randomized controlled experimental design to determine the effect of horticultural practices on internet addiction, social skills and stress levels in children. The children underwent horticultural practices for 6 weeks. Children were given a post-test at the end of the intervention program (week 6), a first follow-up three months after the intervention and a second follow-up six months later.

ELIGIBILITY:
Inclusion Criteria:

* studying in the 6th and 7th grade of secondary school
* volunteering to participate in the research
* consent by the family for participation in the study

Exclusion Criteria:

- the presence of a disease against the materials to be used in horticultural practices (pollen, plant, seed and fertilizer allergy, etc.)

Ages: 11 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Internet Addiction Scale (Internet Addiction Scale for Adolescents) | Baseline (before the intervention)
  The scale consists of nine items. The unidimensional scale has a 5-point Likert-type rating. The responses to the items are graded as 'never', 'rarely', 'sometimes', 'often' and 'always'. The lowest score is 9 points and the highest score is 45 points. The higher the score obtained from the scale, the higher the level of internet addiction.
Social skills scale | 6th week after the intervention
  The Social Skills Scale consists of 20 items. The scale evaluates whether primary and secondary school students display social skill behavior. The response format is a four-point Likert type and consists of the options 1= never, 2= sometimes, 3= usually and 4= completely. The lowest score obtained from the scale is 20, the highest score is 80. A low score from the scale indicates inadequacy in displaying this behavior in terms of social skills, while a high score indicates adequacy in displaying social skill behavior.
Social skills assessment scale | three months after completion of the intervention
  The Social Skills Assessment Scale was developed to measure skills that are important in helping communication deficiencies to increase interaction. The scale is a five-point Likert-type scale and social skills are assessed by families. The skills that children should have in the scale consist of twelve subcategories. The social skills assessment scale is completed by families.
Perceived stress scale in children | six months after completion of the intervention
  The Scale of Perceived Stress in Children was developed by Snoeren-Hoefnagels (2014). The child is asked to answer how appropriate each item is for him/her. The scale consists of 9 items. The one-dimensional scale has a four-point Likert-type rating. High scores from the scale questions mean that the individual's stress level is high.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Emek/Çankaya, Turkey (Türkiye)